CLINICAL TRIAL: NCT04277234
Title: Functional Characterisation of Post-stroke Fatigue: a Cross-sectional Study
Brief Title: Functional Characterisation of Post-stroke Fatigue
Acronym: PSF-SAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Collaborators: Centre Hospitalier Universitaire UCLouvain Namur (Other); CHU Ambroise-Paré - Mons (Unknown)
Responsible Party: Sponsor
Other Study IDs: PSF-SAG; 2017/14SEP/443 (Other: CEHF)
Record Dates: First submitted 2019-02-21; First posted 2020-02-20 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Stroke; Stroke Sequelae
Keywords: fatigue; fatigability; functional impairment
MeSH Terms: conditions — Stroke; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-stroke fatigue is highly prevalent and disabling. However, its causes and consequences in the chronic phase are not fully understood. The aim of this cross-sectional study is to explore functional correlates of post-stroke fatigue in the chronic phase.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Evaluation > 24
* Stroke > 6 months ago

Exclusion Criteria:

* Current active infection
* Multiple stroke
* Other affection of the central nervous system
* Medication potentially inducing severe fatigue
* Hospital admission during last month
* Severe Apraxia
* Severe Aphasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | assessment during 1 day study visit
  9-item fatigue scale (Score/7) Minimum value = 1, Maximum value = 7 An average score greater than or equal to four signifies pathological fatigue

SECONDARY OUTCOMES:
Pittsburgh Sleep quality index | assessment during 1 day study visit
  Sleep assessment. The score of seven components are summed to provide a global score from 0 to 21.
  A global score greater than five is indicative of poor sleep
ACTIVLIM specific to patients with stroke | assessment during 1 day study visit
  Rasch-validated activity assessment. Self-report 20-item questionnaire based on the International Classification of Functioning, Disability and Health and includes activities related to self-care, transfer, mobility, manual ability and balance.
  Participants have to evaluate the perceived difficulty of performing each activity if realised without technical or human assistance. Each item has three response possibilities (impossible, difficult, easy)
Hospital Anxiety and Depression Scale (HADS) | assessment during 1 day study visit
  Mood assessment. Self-report questionnaire with anxiety and depression subscales, each consisting of 7 questions.
  Score each item from 0 (no symptoms) to 3 points (maximum impairment) The cutoff for a pathological score is ≥ 7 for each subscale
6-minute walk test | assessment during 1 day study visit
  Speed decrement (distance first minute - distance last minute). The distance walked each minute and the total distance walked were measured. Performance fatigability was assessed by the difference of distance walked during the first and sixth minutes.
Neuromuscular Fatigability Index | assessment during 1 day study visit
  Decrement in isometric strength of knee extensors during fatiguing task The NMFI is calculated by the difference between the putative torque-versus-time curve if the subject had maintained the maximal torque recorded during the first 5 seconds for 45 seconds, considered as a score of 100 arbitrary units, and the actual area under the torque-versus-time curve.
  A higher NMFI score indicates higher fatigability

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Rahamatali M, De Bont N, Valet M, Halkin V, Hanson P, Deltombe T, Lejeune T, Selves C. Post-stroke fatigue: how it relates to motor fatigability and other modifiable factors in people with chronic stroke. Acta Neurol Belg. 2021 Feb;121(1):181-189. doi: 10.1007/s13760-020-01453-9. Epub 2020 Aug 1. PMID 32740873